CLINICAL TRIAL: NCT05052255
Title: An Open-label, Single Agent, Phase I/II Trial Investigating the Safety and Efficacy of RVU120 (SEL120) in Patients with Relapse / Refractory Metastatic or Advanced Solid Tumors
Brief Title: RVU120 (SEL120) in Patients with Relapse/Refractory Metastatic or Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVU120-SOL-021
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
Keywords: Relapse; Refractory; Metastatic; Advanced; Solid Tumor
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part 1: Dose Escalation / Part 2: Cohort Expansion (Experimental): Part 1-Dose Escalation: Escalating doses of RVU120, in patients who have progressed from previous therapy.
  Part 2-Cohort Expansion and Alternative Schedule Investigation: Recommended dose in patients with tumor types selected from part 1 and escalation for alternative schedule.
  Interventions: Drug: RVU120

INTERVENTIONS:
Drug: RVU120 — RVU120 will be administered as a single oral dose every other day over a 3 week treatment cycle until disease progression or unacceptable toxicity and an alternative daily dosing schedule will also be tested.

SUMMARY:
This is a phase 1/2, dose-escalation and expansion study investigating the safety, pharmacokinetics, and efficacy of RVU120 (SEL120) in patients with metastatic or advanced solid tumors progressing from previous lines of therapy.

DETAILED DESCRIPTION:
The dose-escalation phase (Part 1) will be followed by an expansion phase (Part 2). Part 1 will evaluate the safety/tolerability and pharmacokinetics of increasing doses of RVU120 (SEL120) administered as a single dose every other day (7 doses in a 3 week cycle). Part 2 will collect additional data on safety, pharmacokinetics and efficacy at the recommended dose in patients with tumor types selected in Part 1.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older;
2. Histologically confirmed and/or documented advanced or metastatic tumors who have exhausted the available standard treatment(s) of the respective country and/or progressing from at least one previous systemic therapy and not eligible to further available therapy;
3. At least one measurable or evaluable disease according to RECIST v1.1;
4. Performance status of ECOG 0-2;
5. Estimated life expectancy of at least 12 weeks;
6. Toxicities incurred as a result of previous anti-cancer therapy resolved to ≤ Grade 1 (as defined by NCI CTCAE v5.0), except for alopecia, lymphopenia assessed as non-clinically significant, sensory neurotoxicity and erectile dysfunction that could be ≤ G2;
7. At least a 4-week interval between the last received radiotherapy and the first scheduled day of dosing with RVU120 (SEL120) (with the exception of palliation radiotherapy which is allowed up to 2 weeks prior the first scheduled day of dosing);
8. Complete recovery from major surgery (stable and < Grade 2 toxicity sequela acceptable);
9. At least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids < 20 mg prednisone or equivalent daily are permitted);
10. Laboratory values at Screening and or at D1C1 pre-dose:

    1. Absolute neutrophil count ≥1.5 x 109/L without colony stimulating factor support;
    2. Platelets 100 x 109/L;
    3. Only for Part 1: Hemoglobin ≥9 g/dL (or ≥2.2 mmol/L) without RBC transfusion within 4 weeks;
    4. Serum albumin ≥ 30g/L (3.0g/dL);
    5. Total bilirubin <1.5 times the upper limit of normal (ULN);
    6. AST (SGOT) ≤3 x ULN; ALT (SGPT) ≤3 x ULN; (≤5 x ULN for patients with advanced solid tumors with liver metastases); ALP ≤5 x ULN for patients with advanced solid tumors with bone or liver metastases
    7. Creatinine clearance ≥60 mL/min (Cockroft-Gault formula Appendix 4);
    8. Normal coagulation (elevated INR, prothrombin time or APTT <1.3 x ULN acceptable);
11. Left ventricular ejection fraction> 50% by echocardiogram or MUGA;
12. Able to provide an archival or fresh tumor biopsy sample at Screening. For patients in Part 2 of study, baseline tumor biopsy samples from progressive disease lesions, where feasible, are required;
13. For women of childbearing potential (WOCBP), a negative pregnancy test must be confirmed before enrolment. WOCBP must commit to using highly effective contraception during study participation and until 6 months after the last dose of study drug. Females must also refrain from donating blood or egg (ovum) during the same time-period;
14. For males, an effective barrier method of contraception must be used during study participation until 6 months after the last dose of study drug, if the patient is sexually active with a WOCBP. Males must also refrain from donating blood or sperm during the same time-period;
15. Ability to give written, informed consent prior to any study-specific Screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice;
16. Capable of understanding the mandated and optional protocol requirements, is willing and able to comply with the study protocol procedures and has signed the main informed document prior to any study specific procedure. For any optional biopsy sampling (tissue and/or blood) and long-term sample storage, additional consent is required;
17. Patients must have been off anti-cancer treatment and prohibited concomitant medications, for 4 weeks or 5 half-lives, whichever is shorter;

    Specific Additional Inclusion Criteria for Part 2 (Group A1):
18. Histologically or cytologically confirmed TNBC of the MSL subtype based on the most recent analyzed biopsy or other pathology specimen.

    Specific Additional Inclusion Criteria for Part 2 (Group A2):
19. Histologically or cytologically confirmed TNBC other than the MSL subtype based on the most recent analyzed biopsy or other pathology specimen.

Exclusion Criteria

1. Active brain metastasis [patients with treated, non-progressive brain metastases, off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks can be enrolled in the trial];
2. Prior history of or planned organ or hematopoietic stem cell transplant;
3. Evidence of ongoing and uncontrolled systemic bacterial, fungal, or viral infection and acute inflammatory conditions (including pancreatitis);
4. Known HIV infection with a CD4+ T-cell (CD4+) count of less than 350 cells/μL or a history of AIDS defining opportunistic infection within the past 12 months or on established antiretroviral therapy for less than 4 weeks or presenting with a viral load of more than 400 copies/mL prior to enrollment or on antiretroviral therapy or prophylactic antimicrobials that are expected to cause significant DDIs or overlapping toxicities with study treatment and cannot be changed to alternative agents;
5. Known positive test of / or known active diagnosis of COVID-19 viral infection.
6. Ongoing significant liver disease such as cirrhosis, drug-induced liver injury, active hepatitis or chronic persistent hepatitis B and/or C;

   * Positive serologic or PCR test results for acute or chronic HBV infection. Patients whose HBV infection status cannot be determined by serologic test results must be negative for HBV by PCR to be eligible for study participation. (www.cdc.gov/hepatitis/hbv/pdfs/serologicchartv8.pdf)
   * Acute or chronic HCV infection. Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation.
7. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RVU120 (SEL120) (e.g., active inflammatory bowel disease, ulcerative disease, malabsorption syndrome, short bowel syndrome, uncontrolled nausea, persistent vomiting or diarrhea);
8. Ongoing drug-induced pneumonitis;
9. Concurrent participation in another investigational clinical trial;
10. Taking any medications, herbal supplements or other substances (including smoking) that are known to be strong inhibitors or strong inducers or sensitive substrates of CYP1A2; with the exception of antibiotics, antifungals, and antivirals that are used as the standard of care or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient and no suitable or available alternative could be found, with prior approval of the Sponsor Study Medical Director;
11. Mean measurement QTcF of >470 msec on triplicate electrocardiograms (ECGs) performed within 5 minutes of each other, using QTcF (Fredericia) formulation;
12. Currently taking drugs that are documented in the drug package insert, to have risk of causing prolonged QTc or torsades de pointes (TdP) (unless these can be changed to acceptable alternatives or discontinued). Please also consult the following Credible Meds web page: https://crediblemeds.org/index.php/login/dlcheck (antibiotics, antifungals, and antivirals that are used as standard of care or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient and no suitable or available alternative could be found, can be used with prior approval by Sponsor Study Medical Director)
13. Patients with clinically significant cardiovascular disease. This includes: Myocardial infarction or unstable angina < 6 months prior to Screening; NYHA Grade III or greater congestive heart failure (Appendix 8); cerebrovascular accident including transient ischemic attack within the past 6 months; Uncontrolled hypertension; Serious or uncontrolled cardiac arrhythmia; Personal history of Torsade de Pointe or syndrome of congenital QTc prolongation or QTc > 470 msec.;
14. Any other prior or current medical condition, intercurrent illness, surgical history, physical or electrocardiogram (ECG) findings, laboratory abnormalities, or extenuating circumstance (e.g., alcohol or drug addiction) that, in the Investigator's opinion, could jeopardize patient safety or interfere with the objectives of the study;
15. Pregnant or breast-feeding females;

    Specific Exclusion Criteria for Part 2, Group A1 and A2:
16. Prior history of malignancies other than TNBC, unless the patient has been free of the disease for 5 years or more prior to Screening. Exceptions to the ≥5-year time limit include history of the following:

    1. basal cell carcinoma of the skin;
    2. non-metastatic squamous cell carcinoma of the skin;
    3. carcinoma in situ of the cervix;
    4. carcinoma in situ of the breast;
    5. carcinoma in situ of the bladder;
    6. incidental histological finding of prostate cancer (Tumor/Node/Metastasis [TNM] stage of T1a or T1b).
17. More than 3 prior lines of systemic therapy for metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events in part I | Up to 2 years
  Evaluation of frequency and nature of adverse events, serious adverse events and dose limiting toxicities
Dose Finding in part I | Up to 2 years
  Determination of Recommended phase 2 dose assessing all available data
Objective Overall Response in part II | Up to 2 years
  Objective Overall Response as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (v1.1)
Duration of Response in part II | Up to 2 years
  Duration of Response, as Assessed by RECIST v1.1
Progression Free Survival in part II | Up to 2 years
  Progression Free Survival as Assessed by RECIST v1.1
Overall Survival in part II | Up to 2 years
  Assessment of Overall Survival from the date of first dose until the date of death from any cause

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 2 years
  Assessed of the maximum plasma concentration (Cmax)
Minimum Plasma Concentration (Cmin) | Up to 2 years
  Assessed of the minimum plasma concentration (Cmin)
Time to Cmax | Up to 2 years
  Assessed of the Time to Cmax (Tmax)
Area Under the Curve | Up to 2 years
  Assessed of the Area Under the Concentration Time-Curve (AUC) from Time Zero to Dosing Interval (AUC0-tau)
Objective Overall Response | Up to 2 years
  Objective Overall Response as Assessed by RECIST v1.1
Duration of Response | Up to 2 years
  Duration of Response, as Assessed by RECIST v1.1
Progression Free Survival | Up to 2 years
  Progression Free Survival as Assessed by RECIST v1.1
Overall Survival | Up to 2 years
  Assessment of Overall Survival from the date of first dose until the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (7):
- Poland (4):
  - Beskidzkie Centrum Onkologii, Szpital Miejski im., Bielsko-Biala
  - Medical University Early Phase 1 Research Center / Uniwersyteckie Centrum Kliniczne Ośrodek Badań Klinicznych Wczesnych Faz, Gdansk
  - UCK im. prof. K. Gibińskiego, Katowice
  - Maria Sklodowska-Curie National Research Institute of Oncology / Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Spain (3):
  - Next Oncology Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Next Oncology Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No